CLINICAL TRIAL: NCT01512251
Title: A Phase 1/2 Trial of BKM120 Combined With Vemurafenib (PLX4032) in BRAFV600E/K Mutant Advanced Melanoma (Novartis Study Number CBKM120ZUS21T)
Brief Title: BKM120 Combined With Vemurafenib (PLX4032) in BRAFV600E/K Mutant Advanced Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Alain Algazi, Assistant Clinical Professor - Melanoma Oncology, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11952; CBKM120ZUS21T (Other: Novartis)
Record Dates: First submitted 2011-12-20; First posted 2012-01-19 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: BRAF Mutant Metastatic Melanoma
Keywords: BKM120; BRAF; Melanoma; PI3K
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No Previous Treatment (Other): 150 mg oral dabrafenib twice a day until disease progression, death, or unacceptable adverse events.
  Interventions: Drug: BKM120 Combined with Vemurafenib (PLX4032)

INTERVENTIONS:
Drug: BKM120 Combined with Vemurafenib (PLX4032) — Phase I is 3+3 dose escalation study to identify the recommended phase 2 dose (RP2D)
  Dose Level -1: BKM120 60 mg daily, Vemurafenib 480 mg bid
  Dose Level 1: BKM120 60 mg daily, Vemurafenib 720 mg bid
  Dose Level 2: BKM120 80 mg daiy, Vemurafenib 720 mg bid
  Dose Level 3: BKM120 100 mg daiy, Vemurafenib 720 mg bid
  Dose Level 4: BKM120 100 mg daiy, Vemurafenib 960 mg bid
  Phase II is a single-stage, single arm prospective trial: patients will receive BKM120 and vemurafenib at the RP2D

SUMMARY:
This is a phase 1/2 clinical trial with the goal of determining whether the addition of the investigational agent BKM120 to vemurafenib will lead to improved 6-month progression-free survival in patients with BRAFV600E/K mutant melanoma.

DETAILED DESCRIPTION:
The phase 1 portion of this trial is a dose escalation study; the phase 2 portion is a single-stage, single arm prospective clinical trial. All patients will receive continuous doses of vemurafenib twice a day and BKM120 once a day.

In the phase 1 portion of the study, there will be a 7 day lead-in period to allow for single dose pharmacokinetic analysis of BKM120 alone. Cycle 1 (28 days) is the dose-limiting toxicity (DLT) period. During phase 1, vemurafenib and BKM120 doses will be escalated using a standard 3+3 dose escalation scheme with the goal of identifying the recommended phase 2 dose.

In the phase 2 portion of the study, patients will receive continuous doses of vemurafenib and BKM120 starting on day 1 of the first cycle. In the phase 2 portion of the study, patients will receive vemurafenib and BKM120 at the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed diagnosis of unresectable stage III and stage IV melanoma
2. BRAFV600E or BRAFV600K mutation-positive
3. Age >= 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status <= 2
5. Patients must have at least one site of measurable disease (per RECIST for solid tumors)
6. Life expectancy of ≥ 12 weeks
7. Adequate bone marrow function as shown by: Absolute Neutrophil Count (ANC) >= 1.5 x 109/L, Platelets >= 100 x 109/L, Hb >9 g/dL
8. Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
9. Magnesium ≥ the lower limit of normal
10. Potassium within normal limits for the institution
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or <= 3.0 x upper limit of normal (ULN) if liver metastases are present)
12. Serum bilirubin within normal range (or <= 1.5 x ULN if liver metastases are present; or total bilirubin <= 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
13. Serum creatinine <= 1.5 x ULN or 24-hour clearance >= 50 mL/min
14. Serum amylase <= ULN
15. Serum lipase <= ULN
16. International Normalized Ratio (INR) <= 2
17. Fasting plasma glucose <= 120 mg/dL (6.7 mmol/L)
18. Negative serum pregnancy test within 48 hours before starting study treatment

Exclusion Criteria

1. Patients who have received prior treatment with a PI3K inhibitor or a BRAF inhibitor, prior treatment with sorafenib is permitted.
2. Patients with a known hypersensitivity to BKM120 or to its excipients
3. Patients with untreated brain metastases are excluded; however, patients with metastatic central nervous system (CNS) tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (incl. radiation and/or surgery) and clinically stable at the time of study entry
4. Patients with acute or chronic liver, renal disease or pancreatitis
5. Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire:

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, history of suicidal attempt or ideation, or homicidal ideation
   * >= CTCAE grade 3 anxiety
   * Meets the cut-off score of >= 10 in the Patient Health Questionnaire-9 (PHQ-9) or a cut-off of >= 15 in the General Anxiety Disorder-7 (GAD-7) mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study unless overruled by the psychiatric assessment
6. Patients with diarrhea >= CTCAE grade 2
7. Patient has active cardiac disease including any of the following:

   * Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition (MUGA) or echocardiogram (ECHO)
   * QTc > 480 msec on screening ECG (using the QTcF formula)
   * Personal or family history of prolonged QT syndrome
   * Angina pectoris that requires the use of anti-anginal medication
   * Ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Symptomatic pericarditis
8. Patient has a history of cardiac dysfunction including any of the following:

   * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular ejection fraction (LVEF) function
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
9. Poorly controlled diabetes mellitus (HbA1c > 8 %)
10. Other concurrent severe and/or uncontrolled concomitant medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol

    - Significant symptomatic deterioration of lung function; if clinically indicated, pulmonary function tests including measures of predicted lung volumes, Diffusing capacity of the lungs for carbon monoxide (DLCO), oxygen (O2) saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
11. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
12. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., Granulocyte colony-stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF)) <= 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
13. Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
14. Patients receiving chronic treatment with steroids or another immunosuppressive agent; topical applications, inhaled sprays, eye drops or local injections are allowed; patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment for at least 14 days before start of study treatment are eligible
15. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug - herbal medications include, but are not limited to St. John's Wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; fruits include CYP3A inhibitors: Seville oranges, grapefruit, pomelos, or exotic citrus fruits
16. Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug; note that co-treatment with weak inhibitors of CYP3A is allowed).
17. Patients who have received chemotherapy or targeted anticancer therapy <= 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must have resolution of treatment related adverse events to baseline or grade 1 before starting the trial
18. Patients who have received wide field radiotherapy <= 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
19. Patients who have undergone major surgery <= 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
20. Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant
21. Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control; women of child-bearing potential must have a negative serum pregnancy test <= 72 hours prior to initiating treatment; double barrier contraceptives must be used through the trial by both sexes; oral, implantable, or injectable contraceptives are therefore not considered effective for this study

    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 milli-international units per millilitre (mIU/mL) [for US only: and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
    * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment for 3 months in total after study drug discontinuation. Highly effective contraception is defined as either: True abstinence-when this is in line with the preferred and usual lifestyle of the subject, periodic abstinence and withdrawal are not acceptable methods of contraception; Sterilization-have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; Male partner sterilization-for female subjects, the vasectomised male partner should be the sole partner for that patient; Use of a combination of any two of the following barrier methods of contraception-condom or Occlusive cap with spermicidal foam/gel/film/cream/vaginal suppository
    * Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment, for 3 months in total after study drug discontinuation and should not father a child in this period
22. Known diagnosis of human immunodeficiency virus (HIV) infection
23. History of another malignancy within 3 years, except cured or curable basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix; patients with lesions curable by excision must have these lesions excised prior to the initiation of treatment on study
24. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06-09 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Algazi AP, Rotow J, Posch C, Ortiz-Urda S, Pelayo A, Munster PN, Daud A. A dual pathway inhibition strategy using BKM120 combined with vemurafenib is poorly tolerated in BRAF V600E/K mutant advanced melanoma. Pigment Cell Melanoma Res. 2019 Jul;32(4):603-606. doi: 10.1111/pcmr.12777. Epub 2019 Apr 13. No abstract available. PMID 30801911

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib-Naïve; Vemurafenib-Resistant: 150 mg oral dabrafenib twice a day (bid) until disease progression, death, or unacceptable adverse events.
  Dose Level -1:
  BKM120 60 mg daily Vemurafenib 480 mg bid
  Phase I, Dose Level 1:
  BKM120 60 mg daily Vemurafenib 720 mg bid
  Phase I, Dose Level 2:
  BKM120 80 mg daily Vemurafenib 720 mg bid
  Phase I, Dose Level 3:
  BKM120 100 mg daily Vemurafenib 720 mg bid
  Phase I, Dose Level 4 BKM120 100 mg daily Vemurafenib 960 mg bid
  Phase II 150 mg oral dabrafenib twice a day (bid) until disease progression, death, or unacceptable adverse events.
  BKM120 Combined with Vemurafenib (PLX4032): Phase I is 3+3 dose escalation study to identify the recommended phase 2 dose (RP2D)
Period: Dose Level -1
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Phase I, Dose 1
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Started | 3 | 5
Completed | 0 | 0
Not Completed | 3 | 5
Period: Phase I, Dose 2
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Phase I, Dose 3
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Phase I, Dose 4
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Phase II
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 44 [26 to 75] | 51 [40 to 62] | 50 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Safety & Recommended Phase 2 Dose (RP2D)
Description: RP2D determined by maximum tolerated dose (MTD), post-dose-limiting toxicity (DLT) period toxicity, and pharmacokinetic data
Time Frame: 28 days
Measure: Number; unit: mg
Groups:
- Determination of MTD: Vemurafenib-Naïve and Vemurafenib-Resistant populations received:
  150 mg oral dabrafenib twice a day (bid) until disease progression, death, or unacceptable adverse events.
  Dose Level -1:
  BKM120 60 mg daily Vemurafenib 480 mg bid
  Phase I, Dose Level 1:
  BKM120 60 mg daily Vemurafenib 720 mg bid
Arm/Group | Determination of MTD
Number analyzed (Participants) | 8
mg | 60

2. Primary Outcome: Phase 2 - Progression-free Survival Rate
Description: 6 month progression-free survival rate (PFS6) determined by tumor assessments, clinical tests and laboratory tests
Time Frame: 6 months
Population: Data were not collected, study never advanced to Phase II.
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Secondary Outcome 1 Phase 2 - Objective Response Rate
Description: Objective response rate determined by tumor assessments, clinical tests and laboratory tests.
Time Frame: Day 28 (+/- 3) of even-numbered treatment cycles until progression
Population: Data not collected
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Secondary Outcome 2 Phase 2 - Safety and Tolerability
Description: Determined by clinical and laboratory tests, and adverse events (AE) assessments
Time Frame: During study treatment, up to 2 years
Population: Data not collected
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Secondary Outcome 3 Phase 2 - Phosphatase and TENsin (PTEN) Expression
Description: PTEN expression associated with better PFS determined by laboratory tests.
Time Frame: No time limit
Population: Data not collected
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Secondary Outcome 4 Phase 2 - Phosphatidylinositol 3-kinase (PI3K)-Pathway Signaling Reduction Levels
Description: Greater reduction in PI3K-pathway signaling associated with better PFS determined by laboratory tests and tumor assessments.
Time Frame: No time limit
Population: Data not collected: study was terminated early due to dose limiting toxicities.
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Secondary Outcome 5 Phase 2 - PI3K Pathway Gene Expression Levels
Description: Responding tumors lack gene expression signatures of PI3K pathway activation, and progressing tumors demonstrate gene expression signatures of PI3K pathway activation - determined by laboratory tests and tumor assessments.
Time Frame: No time limit
Population: Data not collected
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Secondary Outcome 6 Phase 2 - MAPK Pathway Gene Expression Levels
Description: Responding tumors lack gene expression signatures of MAPK pathway activation, and progressing tumors demonstrate gene expression signatures of MAPK pathway activation - determined by laboratory tests and tumor assessments.
Time Frame: No time limit
Population: Data not collected
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vemurafenib-Naïve | Vemurafenib-Resistant
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib-Naïve (N=3) | Vemurafenib-Resistant (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Biliary Fistula (Hepatobiliary disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Renal insufficiency (Blood and lymphatic system disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib-Naïve (N=3) | Vemurafenib-Resistant (N=5)
elevated LDH (Blood and lymphatic system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
adrenal insufficiency (Endocrine disorders) | 1 | 0
eye redness (Eye disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 1
vomiting (Gastrointestinal disorders) | 1 | 2
diarrhea (Gastrointestinal disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Chills (General disorders) | 1 | 1
fatigue (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Rash on lower abdomen (Infections and infestations) | 0 | 1
MRSA infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
weight loss (Investigations) | 2 | 0
QtC Prolongation (Investigations) | 1 | 0
creatinine increased (Investigations) | 1 | 0
alkaline phosphatase increased (Investigations) | 1 | 0
ALT increased (Investigations) | 1 | 0
AST increased (Investigations) | 1 | 0
Decreased wbc (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
hypokalemia (Metabolism and nutrition disorders) | 1 | 0
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
hyponatremia (Metabolism and nutrition disorders) | 2 | 0
hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
anorexia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint pain (pain in extremity) (Musculoskeletal and connective tissue disorders) | 0 | 1
fingertip numbness (Nervous system disorders) | 1 | 0
headache (Nervous system disorders) | 1 | 0
Restlessness (Nervous system disorders) | 0 | 1
Tingling Extremities (Parasthesia) (Nervous system disorders) | 0 | 1
somnolence (Nervous system disorders) | 1 | 0
tremor (Nervous system disorders) | 1 | 0
anxiety (Psychiatric disorders) | 1 | 0
depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Decreased concentration (Psychiatric disorders) | 1 | 0
proteinuria (Renal and urinary disorders) | 1 | 0
Groin/testicular pain (Reproductive system and breast disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinnorhea (Pharyngeal mucositis) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 3 | 1
photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
desquamation of hands & feet (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Crust on elbow (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythemia nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Decreased activity level (General disorders) | 1 | 0
high eosinophil count (Blood and lymphatic system disorders) | 1 | 0
LDH increased (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
low hematocrit (Blood and lymphatic system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to dose limiting toxicities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-06-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT01512251/Prot_SAP_000.pdf
  • Informed Consent Form (2013-06-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT01512251/ICF_001.pdf